CLINICAL TRIAL: NCT01084759
Title: A Pilot Study of Parenteral Testosterone and Oral Etoposide as Therapy for Men With Castration Resistant Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J09121, NA_00033419
Record Dates: First submitted 2010-03-09; First posted 2010-03-10 (Estimated); Results first posted 2016-05-09 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Testosterone; testosterone 17 beta-cypionate; Etoposide; etoposide phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Etoposide and Testosterone (Experimental): Patients will receive an intramuscular gluteal injection with testosterone cypionate at a dose of 400 mg every month for a total of 3 injections (i.e. 3 months of therapy).On the day of testosterone injection (i.e. day 1 of each cycle) patients will begin therapy with oral etoposide at a dose of 100 mg/day given in divided doses (one 50 mg etoposide capsule q 12 h) for 14 consecutive days.
  Interventions: Drug: Testosterone injection; Drug: Etoposide

INTERVENTIONS:
Drug: Testosterone injection — Patients will receive an intramuscular gluteal injection with testosterone cypionate at a dose of 400 mg every month for a total of 3 injections (i.e. 3 months of therapy). This route and dose of testosterone was selected based on data demonstrating that it produces an initial supraphysiologic serum level of testosterone (i.e. > 3-5 times normal level) with eugonadal levels achieved at the end of two weeks.
  Other Names: Testosterone Cypionate
Drug: Etoposide — On the day of testosterone injection (i.e. day 1 of each cycle) patients will begin therapy with oral etoposide at a dose of 100 mg/day given in divided doses (one 50 mg etoposide capsule q 12 h) for 14 consecutive days. This dose was selected based on Phase II studies of the combination of oral estramustine and oral etoposide. In these trials, myelosuppression was observed when etoposide was given for 21 days out of a 28 day cycle. Therefore, to minimize toxicity, in this study etoposide will be administered for 14 days of a 28 day cycle.
  Other Names: Etopophos; Toposar

SUMMARY:
The objective of the study is to determine if men with evidence of progressive prostate cancer while on chronic androgen ablation of ≥ 1 year duration will exhibit a clinical response following administration of parenteral testosterone and oral etoposide.

Treatment Plan: Eligible patients will continue on androgen ablative therapy with luteinizing hormone-releasing hormone (LHRH) agonist (i.e. Zoladex or Lupron) if not surgically castrated. Patients will receive intramuscular injection with testosterone cypionate at a dose of 400 mg every month for a total of 3 injections (i.e. 3 months of therapy). This dose was selected based on data demonstrating that it produces an initial supraphysiologic serum level of testosterone (i.e. > 3-5 times normal level) with eugonadal levels achieved at the end of two weeks. Beginning the day of the testosterone injection, patients will also receive oral etoposide 100 mg/day in divided doses (50 mg q 12h) x 14 days out of 28 days per cycle. After 3 months on therapy, patients will have repeat prostate specific antigen (PSA) and bone/computed tomography (CT) scans to establish the effect of combined testosterone and etoposide treatment on these parameters (i.e. "testosterone effect baseline"). Patients with sustained elevations in PSA ≥ 50% above pre-testosterone treatment PSA levels after the initial three months of testosterone and etoposide therapy will not receive continued therapy and will come off study. Patients with PSA levels less than the peak serum PSA level seen over the three month period (PSA decline) or patients with PSA ≤ 50% of pretreatment baseline will receive a second 3 month course of monthly testosterone and etoposide therapy until evidence of disease progression. Disease progression is defined as a PSA increase above the PSA level obtained after 3 months on testosterone treatment over two successive measurements 2 weeks apart or evidence of new lesions or progression on bone/CT scans compared to baseline studies. Patients who respond to initial treatment with testosterone and etoposide and then show signs of progression will have the option of retreatment with testosterone alone after a period of 3 months or greater off of the original therapy.

DETAILED DESCRIPTION:
Based on our preclinical data, high levels of androgens can lead to significant growth suppressive effects in prostate cancer cells in vitro and in vivo. Mechanistic data in in vitro models suggests that this growth suppression may be due to the accumulation of androgen induced TOP2B mediated double strand breaks at AR target sites occurring after stimulation of prostate cancer cells with high levels of androgens. Provocatively, the number of double strand breaks was significantly increased (Figure 3 B) if the cells were treated with etoposide, an agent that leads to formation of double strand breaks at TOP2 target sites, concurrently with high-dose androgen stimulation. We hypothesize that co-administration of testosterone with etoposide could produce high levels of double strand breaks in prostate cancer cells, overwhelming DNA repair and survival mechanisms and leading to cancer cell death or growth arrest. To test whether this possibility holds promise for therapy of advanced prostate cancer, we propose the following clinical trial of parenteral testosterone therapy in combination with oral etoposide in men with evidence of progressive prostate cancer during chronic androgen ablation.

ELIGIBILITY:
Inclusion Criteria:

1. Performance status ≤2
2. Documented adenocarcinoma of the prostate with histologic confirmation
3. Treated with continuous androgen ablative therapy (either surgical castration or LHRH agonist for ≥ 1 year)
4. Documented castrate level of serum testosterone (<50 ng/dl)
5. Evidence of rising PSA on two successive dates > 1 month apart
6. Treatment with ≤ 2 prior chemotherapeutic regimens allowed
7. Treatment with ≤2 prior second line hormone therapies allowed.
8. Prior treatment with ketoconazole is allowed.
9. Patients must be withdrawn from antiandrogens for ≥ 6 weeks and have documented PSA increase after the 6 week withdrawal period.
10. Patients with rising PSA only or ≤ 5 sites of asymptomatic bone metastases and < 10 total sites of disease including bone and soft tissue documented within 28 days of enrollment on trial.
11. Patients will considered for repeat treatment with testosterone if they meet the following criteria:

    1. Had either PSA decline from baseline following treatment with testosterone or had return of PSA levels to pretreatment baseline once serum testosterone reached a castrate level.
    2. Must continue to meet inclusion/exclusion criteria as described above
    3. Must have been off testosterone therapy for ≥ 3 months
    4. Must have castrate level of serum testosterone
    5. Must have evidence of rising PSA on two occasions at least 2 weeks apart
    6. Are allowed to have had additional treatment with up to 2 additional hormonal therapies that include anti-androgens (e.g. flutamide, bicalutamide, nilutamide, enzalutamide), CYP17 inhibitors (e.g. ketoconazole, abiraterone acetate) or other investigational hormonal therapies.

Exclusion Criteria:

1. Evidence of disease in sites or extent that, in the opinion of the investigator, would put the patient at risk from therapy with testosterone (e.g. femoral metastases with concern over fracture risk, spinal metastases with concern over spinal cord compression, lymph node disease with concern for ureteral obstruction)
2. Abnormal liver function (bilirubin, AST, ALT ≥ 2 x upper limit of normal)
3. Abnormal kidney function (serum creatinine ≥ 2 x upper limit of normal)
4. Inability to provide informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Denmeade, MD, Principal Investigator — Johns Hopkins School of Medicine - Sidney Kimmel Comprehensive Cancer Center; Alberto J Pacheco, BA, Study Chair — Johns Hopkins School of Medicine - Sidney Kimmel Comprehensive Cancer Center; Ting Wang, MS, Study Director — Johns Hopkins School of Medicine - Sidney Kimmel Comprehensive Cancer Center
Locations (1):
- Johns Hopkins School of Medicine - Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Testosterone: Men with castration-resistant prostate cancer will continue on androgen ablative therapy with LHRH agonist (i.e. Zoladex or Lupron) if not surgically castrated. Patients will receive intramuscular injection with testosterone cypionate at a dose of 400 mg every month for a total of 3 injections (i.e. 3 months of therapy).
Period: Overall Study
Arm/Group | Testosterone
Started | 16
Completed | 14
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Etoposide and Testosterone
Number analyzed (Participants) | 16
Age, Continuous [Median (Full Range); unit: years] | 71 [56 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Prostate Specific Antigen (PSA) [Median (Full Range); unit: ng/mL] | 20 [1.4 to 819.1]
Testosterone [Median (Full Range); unit: ng/dL] — Note: The limit of detection for this assay is 20 ng/dL. Patients with an undetectable testosterone level were assigned a value of 20 ng/dL.
  ng/dL | 20 [20 to 41]
Baseline Gleason Grade (higher grade indicates more pathologic atypia) [Number; unit: participants] — Gleason score was based on clinical interpretation of the needle biopsy specimen or prostatectomy specimen by an expert pathologist.
  participants
    Gleason score 6 | 4
    Gleason score 7 | 7
    Gleason score 8 | 3
    Gleason score 9 | 2
Length of continuous androgen deprivation therapy [Median (Full Range); unit: months] | 45.5 [12 to 146]
Number of second line hormonal therapies received [Number; unit: participants] — Second line hormonal therapies were defined as any agent that inhibits androgen receptor (AR) signaling (e.g. AR antagonist, inhibitors of extragonadal testosterone synthesis).
  participants
    None | 2
    1 second line agent | 9
    2 second line agents | 3
    3 second line agents | 2
Bone metastases [Number; unit: participants]
  Patients with bone metastases | 3
  Patients without bone metastases | 13
RECIST evaluable soft tissue metastases [Number; unit: participants]
  Patients with RECIST evaluable disease | 10
  Patients without RECIST evaluable disease | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Completing at Least 3 Months of Therapy With a PSA Below Baseline.
Time Frame: 3 months
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Treatment Group: Testosterone cypionate 400 mg intramuscular, day 1 of 28; etoposide 100 mg oral daily, days 1-14 of 28. Note: Etoposide is only given for 3, 28-day cycles.
Arm/Group | Treatment Group
Number analyzed (Participants) | 14
Percentage of Participants | 42.9 [20.6 to 68.8]

2. Primary Outcome: Time to PSA Progression
Description: Time to a PSA increase above the PSA level obtained after 3 months on testosterone treatment over two successive measurements 2 weeks apart.
Time Frame: 2 years
Measure: Median (Full Range); unit: days
Arm/Group | Treatment Group
Number analyzed (Participants) | 14
days | 221 [95 to 454]

3. Secondary Outcome: Number of Participants With RECIST Response (i.e. Complete Response or Partial Response)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT scan or MRI. Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 14
participants | 7

ADVERSE EVENTS:
Time Frame: 3 years
Groups:
- Treatment Group: Men with castration-resistant prostate cancer will continue on androgen ablative therapy with LHRH agonist (i.e. Zoladex or Lupron) if not surgically castrated. Patients will receive intramuscular injection with testosterone cypionate at a dose of 400 mg every month for a total of 3 injections (i.e. 3 months of therapy).
Arm/Group | Treatment Group
Serious Adverse Events (participants affected / at risk) | 3/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group (N=16)
Pulmonary embolus (Respiratory, thoracic and mediastinal disorders) | 2
Neutropenic fever (Infections and infestations) | 1 — Patient died as a result
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group (N=16)
Nausea (Gastrointestinal disorders) | 10
Fatigue (Nervous system disorders) | 9
Alopecia (Skin and subcutaneous tissue disorders) | 9
Edema (Blood and lymphatic system disorders) | 8
Anemia (Blood and lymphatic system disorders) | 2
Priapism (Reproductive system and breast disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No